CLINICAL TRIAL: NCT06032416
Title: Collection of CT Images to Evaluate Bone Quality Before Total Shoulder Arthroplasty
Brief Title: DenCT Shoulder Bone Quality Evaluation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Zimmer Biomet (Industry)
Collaborators: Zimmer, GmbH (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CSG2023-05E
Record Dates: First submitted 2023-09-04; First posted 2023-09-13 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Osteoarthritis Shoulder; Rotator Cuff Tears
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Shoulder Arthroplasty (Other): Patients in need of a shoulder arthroplasty
  Interventions: Radiation: Preoperative CT Scan

INTERVENTIONS:
Radiation: Preoperative CT Scan — Preoperative CT Scan including a bone density calibration phantom. This data will be compared with surgeon intra-operative CRF responses.

SUMMARY:
The objective of the study is to evaluate the preoperative bone quality assessment based on CT to later establish a scale for the decision of stemless shoulder arthroplasty.

DETAILED DESCRIPTION:
The primary endpoint is the collection of the preoperative CT scan with a calibration phantom at each site and the surgeon's intraoperative evaluation of bone quality. Therefore, this study is not centered around a specific device and any primary shoulder arthroplasty system from Zimmer Biomet including anatomical, hemi, or reverse, stemmed or stemless configurations can be used for the target population. The indications of this study are the shoulder joint diseases such as osteoarthritis and the irreparable rotator cuff tears which are needed with TSA/RSA. The subjects should be also met the inclusion/exclusion criteria. The safety of the system will be assessed by monitoring the frequency and incidence of adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be older than 18 years and skeletally mature.
* Patient must undergo the SHA, TSA, or RSA according to the Instructions for Use (IFU).
* Patient must be anatomically and structurally suited to receive shoulder arthroplasty implants.
* Patient is a candidate for lateral or bi-lateral shoulder arthroplasty due to one or more of the following:
* Non-inflammatory degenerative joint disease including osteoarthritis.
* Avascular necrosis of the humeral head.
* Autoimmune disease including rheumatoid arthritis.
* Irreparable rotator cuff tears.
* Correction of functional deformity.
* Patient must be able and willing to sign the IRB/EC approved informed consent.
* Patient must be able to undergo a preoperative CT scan
* Patient must be willing to share their CT images with sponsor

Exclusion Criteria:

* Patient is a candidate for shoulder arthroplasty due to one or more of the following:
* Fractures of the proximal humerus, where other methods of treatment are deemed inadequate.
* Revision TSA/RSA after the prior TSA/RSA.
* Patient has experienced the traumatic fractures to the implant site.
* Patient is unwilling or unable to give consent
* Patient has any condition which would in the judgement of the Investigator, place the patient at undue risk or interfere with the study, e.g., any neuromuscular disease compromising the affected limb.
* Patient is known to be pregnant or breastfeeding.
* Patient is a vulnerable subject (prisoner, mentally incompetent or unable to understand what participation to the study entails, a known alcohol or drug abuser, and/or anticipated to be non- compliant).
* Patient is uncooperative or patient with neurologic disorders who is incapable or unwilling to follow directions.
* Patient has any sign of infection affecting the shoulder joint or in its proximity which may spread to the implant site.
* Patient has rapid joint destruction, marked bone loss, or bone resorption apparent on roentgenogram.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
CT scan data acquisition | Immediate post-op
  The primary endpoint is the collection of the preoperative CT scan with a calibration phantom at each site and the surgeon's intraoperative evaluation of bone quality.
Intra-op bone quality evaluation: Thumb Test | Intra-op
  The first test is the Thumb test that occurs just after the head resection. The surgeon presses his/her thumb on the resected humeral surface to assess bone quality. If he can depress the thumb into the humerus without much resistance, then primary stability of the stemless implant may be insufficient.
Intra-op bone quality evaluation: Pin Test | Intra-op
  The second test is the Pin test where the central pin used to position the trial head is wiggled to assess bone quality. If the central pin is unstable in the humerus, then this may indicate that the bone is soft/weak.
Intra-op bone quality evaluation: Broach Test | Intra-op
  The third test is the Broach (or Puncher test) where the impactor is wiggled to assess bone quality. If the puncher is unstable after impaction, then the bone is soft/weak, and a stemmed prosthesis is recommended.
Duplicate CT scan data acquisition (Optional) | Immediate post-op
  Additional primary endpoint for a sub-cohort of a maximum of 30 patients. These patients will receive a second preoperative CT scan after a changing position (patient repositioning), which is needed to evaluate the precision of the phantom-less method. This duplicated scan is considered optional in the study.

OTHER OUTCOMES:
Functional Performance (Optional): Constant & Murley Score | Pre-op
  The Constant & Murley Score (CMS) is a multi-item functional scale assessing pain, ADL, ROM and strength of the affected shoulder. Its score ranges from 0 to 100 points, representing worst and best shoulder function, respectively.

CONTACTS AND LOCATIONS:
Overall Officials: Elliott Goff, PhD, Study Chair — Zimmer, GmbH
Locations (1):
- Joint Surgery, Sports Clinic Ishinomaki, Ishinomaki, Miyagi, Japan

IPD SHARING:
Plan to Share IPD: No